CLINICAL TRIAL: NCT05991635
Title: Evaluation of a Gatekeeper Training for Pharmacists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2022-0598
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants in this group (all participants) are asked to complete a questionnaire and then receive access to the online gatekeeper training (e-learning) during three days, after which they were asked to complete another questionnaire. After three months, a third questionnaire is sent.
  Interventions: Behavioral: Gatekeeper training (e-learning)

INTERVENTIONS:
Behavioral: Gatekeeper training (e-learning) — The gatekeeper training consists of an interactive e-learning (min. 1h, max. 3h) which includes theoretical knowledge, tips, exercises and relevant examples and cases. The main topics included in the e-learning are:
  * Background information on suicide in Flanders (rates)
  * Definitions and theoretical background (suicidal process, integrative explanatory model of suicide)
  * Debunking existing myths about suicide
  * The role of the pharmacist in suicide prevention
  * Signal Recognition
  * Talking about suicide and suicidal thoughts (start the conversation)
  * How and to whom to refer as pharmacist or FTA
  * Medication management and medication in the context of suicide
  * Rights and obligations of a pharmacist/PTA in the context of suicide prevention
  * Self-care

SUMMARY:
This study aims to investigate to what extent a gatekeeper training (e-learning) for pharmacists and PTA is effective in changing the attitudes, knowledge, and self-efficacy. Moreover, it aims to examine how they evaluate the training and whether they were able to apply the learned skills in practice.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Have access to internet
* Speak Dutch
* Working as a (public) pharmacist or pharmaceutical technical assistant (FTA)

Exclusion Criteria:

* Hospital pharmacists or industrial pharmacists are not included in this study and thus constitute an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Changes in attitudes: Attitudes Towards Suicide Scale (ATTS) | Change from Baseline (before intervention) to post-test (after a week of access to e-learning)
  The ATTS is a 37-item to be scored on a 5-point Likert scale (1= disagree completely to 5 = agree completely) to measure participants' attitudes towards suicide.

SECONDARY OUTCOMES:
Changes in self-efficacy: Measurement of Perceived Self-efficacy | Change from Baseline (before intervention) to post-test (after a week of access to e-learning)
  The Measurement of Perceived Self-efficacy is a 10-item self-report questionnaire to be scored on a 4-point Likert scale (1= Completely false to 4 = completely true)
Changes in perceptions/myths | Change from Baseline (before intervention) to post-test (after a week of access to e-learning)
  Self-developped questionnaire: 4 statements to be rated as true or false; 2 question about how participant would feel if a patient said they have suicidal thouhgts
Gatekeeper training evaluation | Post-test (after a week of access to e-learning)
  8 evaluative statements about the e-learning to be rated on a 5-point Likert scale (Totally disagree, disagree, neutral, agree, totally disagree).
  Question to rate the e-learning on a scale of 1 (not good at all) to 10 (excellent) Additionally three open questions where participants can give feedback about what they liked/did not like/ general comments.

OTHER OUTCOMES:
Socio-demographic characteristics | Baseline
  Age, Gender, Years of work experience
Previous experience with suicide (prevention) | Baseline and post-test (after a week of access to e-learning)
  At baseline: motivation to participate (9 options), previous trainings (yes/no, specify if yes) At baseline and post-test: experience with suicidal patients (contact and confidence; 5 point Likert scale), knowing what to do or who to refer to (5-point Likert scale), knowing where to find information (5-point Likert scale), which actions previously taken in case of suicidal patient (list of 12), to who do you refer (5 options)
Follow-up | Follow-up (three months after baseline)
  Questions concerning: application of acquired skills and knowledge; actions undertaken in context of suicide prevention (12 options); experienced barriers to application of acquired skills and knowledge; need of extra support

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Phd, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No